CLINICAL TRIAL: NCT05961696
Title: A Phase I Study of Mosunetuzumab for Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0 accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0530; NCI-2023-05744 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Refractory B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mosunetuzumab (Experimental): Participants will be assigned to a dose level of mosunetuzumab based on when the participants join this study. Up to 2 dose levels of mosunetuzumab will be tested. The first group of participants will receive the lowest dose level. A second group will receive a higher dose than the group before it, if no intolerable side effects were seen.
  Interventions: Drug: Mosunetuzumab

INTERVENTIONS:
Drug: Mosunetuzumab — Subcutaneous (SQ or Sub-Q) injection under the skin
  Other Names: RO7030816

SUMMARY:
To find a recommended dose of mosunetuzumab that can be given to patients with ALL.

DETAILED DESCRIPTION:
Primary Objectives:

--To assess the safety of mosunetuzumab in patients with R/R B-ALL

Secondary Objectives:

--To assess rate of CR/CRi, duration of response (DOR), progression-free survival (PFS) and overall survival (OS) of mosunetuzumab in patients with R/R B-ALL

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Signed Informed Consent Form
2. Age 18 years at the time of signing Informed Consent Form
3. Ability to comply with the study protocol
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
5. Histologically confirmed relpased and/or refractory B-ALL with ≥5% marrow blasts or marrow MRD+ (≥0.1%) disease. At least 50% of the blasts must express CD20. Relapsed disease is defined as disease relapse after achieving an initial response to prior therapies. For patients in 1st relapse of their disease, those with CR1 duration >12 months are excluded. Refractory disease is defined as disease refractory to the last therapy received. All patients must have failed or ineligible to receive all therapies with clinical benefit.
6. Adequate organ function:

   * Measured or estimated creatinine clearance 50 mL/min by institutional standard method
   * AST or ALT 2.5 the upper limit of normal (ULN)
   * Serum total bilirubin 1.5 ULN (or 3 ULN for patients with Gilbert syndrome)
   * Ejection fraction ≥50%
7. Adequate BM function independent of growth factor or transfusion support, within 2 weeks of screening, unless cytopenia is clearly due to marrow involvement of B-ALL:

   * Platelet count ≥50,000/mm3
   * ANC ≥500/mm3
   * Hemoglobin ≥9 g/dL
8. WBC ≤10 K/µL at Cycle 1 Day 1
9. For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use 2 adequate methods of contraception, including at least 1 method with a failure rate of 1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period (including periods of treatment interruption), 90 days after the final dose mosunetuzumab. Women must refrain from donating eggs during this same period.

   A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state ( 24 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Even in presence of infertility history, a reliable contraception, including 2 adequate methods of contraception, is indicated.

   Examples of non-hormonal contraceptive methods with a failure rate of 1% per year include bilateral tubal ligation, male sterilization, established and proper use of progestogen only hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices, and copper intrauterine devices. Barrier methods must always be supplemented with the use of a spermicide.
10. For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

    With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 90 days after the final dose of mosunetuzumab. Men must refrain from donating sperm during this same period.

    Exclusion Criteria:

    Patients who meet any of the following criteria will be excluded from study entry:
11. Active CNS disease. Previous history of CNS disease is allowed as long as last documented CNS positivity is >3 months ago, and the last 2 LP are negative for CNS leukemia.
12. Prior standard or investigational anti cancer therapy as specified below:

    * Chimeric antigen receptor T cell therapy within 30 days prior to Day 1 of Cycle 1
    * Monoclonal antibody or antibody drug conjugate within 4 weeks prior to Cycle 1 Day 1
    * Treatment with any anti cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first dose of study treatment
    * Note: For urgent cytoreduction, steroids and hydroxyurea are permitted up to 2 days prior to Cycle 1 Day 1.
13. Clinically significant toxicity (other than alopecia) from prior treatment that has not resolved to Grade 1 (per NCI CTCAE, v5.0) prior to Day 1 of Cycle 1
14. Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone ( 20 mg) within 2 weeks prior to Day 1 of Cycle 1

    * The use of inhaled corticosteroids is permitted
    * The use of mineralocorticoids for management of orthostatic hypotension is permitted
    * Single dose of dexamethasone for nausea or B symptoms is permitted
    * Use of steroids for cytoreduction is permitted as per criteria above
15. History of solid organ transplantation
16. History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies (MAbs)
17. Known hypersensitivity to biopharmaceuticals produced in CHO cells or any component of the mosunetuzumab, lenalidomide, or thalidomide formulation, including mannitol
18. History of erythema multiforme, Grade 3 rash, or blistering following prior treatment with immunomodulatory derivatives
19. Active uncontrolled bacterial, viral, fungal, or other infection
20. Known or suspected chronic active Epstein-Barr virus (EBV) infection
21. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
22. Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
23. Active Hepatitis B infection

    - Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive, must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation
24. Active Hepatitis C infection

    - Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
25. Known history of human immunodeficiency virus (HIV) positive status

    - For patients with unknown HIV status, HIV testing will be performed at screening if required by local regulations
26. History of progressive multifocal leukoencephalopathy (PML)
27. Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment
28. Other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following:

    * Any of the following malignancies previously curatively treated: carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal, or squamous cell skin cancer
    * Stage I melanoma, low grade, early stage localized prostate cancer, or any other previously treated malignancy that has been in remission without treatment for 2 years prior to enrollment
29. Active autoimmune disease requiring treatment
30. History of autoimmune disease, including, but not limited to: myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

    * Patients with a remote history of, or well-controlled autoimmune disease, with a treatment free interval from immunosuppressive therapy for 12 months may be eligible to enroll if judged to be safe by the investigator
    * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone are eligible
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    * Patients with a history of disease-related immune thrombocytopenic purpura, or autoimmune hemolytic anemia may be eligible
31. Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
32. Major surgical procedure within 28 days prior to Day 1 of Cycle 1
33. Pregnant or lactating or intending to become pregnant during the study Women of childbearing potential must have negative serum/urine pregnancy test within 14 days prior to initiating therapy
34. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org